CLINICAL TRIAL: NCT07152132
Title: Slow Coagulation Trans-Scleral Cyclophotocoagulation Versus Trabeculectomy in Medically Uncontrolled Open-Angle Glaucoma in Pseudophakic Patients
Brief Title: SCTSC Versus Trabeculectomy in Medically Uncontrolled Open-Angle Glaucoma in Pseudophakic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hazem Mohamed Mohamed, Assisstant lecture, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SC-TSCPC, Trabeculectomy; SC-TSCPC versus Trabeculectomy (Other: SC-TSCPC versus Trabeculectomy)
Record Dates: First submitted 2025-08-07; First posted 2025-09-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open Angle
Keywords: SC-TSCPC; Trabeculectomy; OAG; Pseudophakic
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 patients will undergo trabeculectomy with MMC (group B). (Active Comparator): 25 patients will undergo trabeculectomy with MMC (group B).
  Interventions: Procedure: Trabeculectomy
- 25 patients will be subjected to SC-TSCPC (group A) (Active Comparator): 25 patients will be subjected to SC-TSCPC (group A)
  Interventions: Procedure: Slow coagulation trans-scleral cyclophotocoagulation

INTERVENTIONS:
Procedure: Trabeculectomy — Trabeculectomy with mitomycin c application
  Arms: 25 patients will undergo trabeculectomy with MMC (group B).
Procedure: Slow coagulation trans-scleral cyclophotocoagulation — Slow coagulation trans-scleral cyclophotocoagulation
  Arms: 25 patients will be subjected to SC-TSCPC (group A)

SUMMARY:
cyclodiode versus trabeculectomy with MMC in pseudophakic patients.

DETAILED DESCRIPTION:
Glaucoma is an optic neuropathy that is characterized by progressive structural and functional neuropathy. It is a leading cause of irreversible blindness.

Open angle glaucoma (OAG) is the commonest subtype of glaucoma. The number of patients diagnosed with POAG was estimated 52.68 million in 2020 and expected to be 79.76 million in 2040.

The management of OAG in patients with pseudophakia aims to IOP, which is the major modifiable risk factor for glaucoma progression. This can be achieved by medical, laser or surgical methods.

In many cases medical therapy can provide an effective IOP control, while surgery and laser are still indicated when the medical treatment fails to lower IOP sufficiently, or if the patient is not compliant with treatment.

Trabeculectomy with mitomycin C (MMC) is a filtration procedure that reduces IOP by creating a connection between the anterior chamber and the sub-conjunctival space after excision of a part of the trabecular meshwork. Pseudophakic eyes with OAG have a higher risk for surgical failure of trabeculectomy with MMC than the phakic eyes. Also it is associated with a higher incidence of complications as hypotony, lost anterior chamber or supra-choroidal effusion.

Laser therapy, as a cyclodestructive procedure, lowers IOP by reducing aqueous humor production. This is achieved through the application of diode laser energy to the sclera, which is absorbed by the melanin pigment in the ciliary processes, resulting in coagulative necrosis of the ciliary body. Historically, this treatment was regarded as a last-resort option for eyes with very limited visual potential due to the significant risks of uncontrolled inflammation and phthisis bulbi.

Now, with recent advances in laser probes and laser settings, the safety of trans-scleral cyclo-destruction has improved, rendering it a viable non-invasive option for a broader spectrum of patients including those with good visual acuity (VA) and as a primary procedure in management of OAG with pseudophakia.

Two approaches are commonly used to deliver laser energy using continuous wave trans-scleral cyclo-photocoagulation (CW-TSCPC): the conventional "pop" technique, where laser energy is initially increased until an audible, explosive, cavitating tissue-derived "pop" is heard. The laser power is then reduced until these pops are no longer audible. This method typically begins with a laser energy setting of approximately 1750-2000 mW, applied for a short duration of 2 seconds, and the treatment is delivered circumferentially along the limbus. In contrast, slow coagulation (SC) CW-TSCPC utilizes a lower amount of diode laser energy over an extended period, approximately 1250 mW over 4 seconds.

Previous results comparing the outcomes of the slow coagulation approach with the conventional high-energy pop approach found a lower incidence of postoperative complications in the slow coagulation group and comparable IOP- lowering effects between both groups. Although conventional CPC may have previously been reserved for blind painful eyes or eyes which have already failed prior glaucoma surgery, recent literature supports slow coagulation TSCPC (SC-TSCPC) as a reasonable primary option to lower IOP in eyes without prior incisional glaucoma surgery.

There have been few reports of SC-TSCPC being used as a primary surgical treatment in patients with glaucoma, and few studies published in the literature documenting the effect of SC-TSCPC in patients with good VA.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients above 40 years old.

  2. POAG who underwent previous uncomplicated cataract surgery with intraocular lens implantation.

  3. Pseudophakic patients with medically uncontrolled glaucoma in spite of the use of two anti-glaucoma medications or intolerance to medical therapy.

  4. Visual field defects in both the superior and inferior hemi-fields outside the central 5 degrees of fixation.

  5. Mean deviation on perimetry ranges between -6 dB and -12 dB

Exclusion Criteria:

* 1. Patients with history of previous glaucoma surgery. 2. Patients who have used topical steroids within the last three months. 3. Patients with significant media opacity, such as corneal opacity, that obstructs fundoscopic examination.

  4. Patients with ocular diseases as uveitis. 5. Patients with severe ocular surface disorders as ocular cicatricial pemphigoid.

  6. Aphakic patients. 7. Ocular interventions apart from YAG posterior capsulotomy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluate and compare the amount of iop reduction between SC-TSCPC and trabeculectomy with MMC in the management of medically uncontrolled OAG in pseudophakic eyes. | 6 months
  measuring the IOP with Goldman applanation tonometer.
evaluate and compare the degree of safety of SC-TSCPC versus trabeculectomy with MMC in the management of medically uncontrolled OAG in pseudophakic eyes. | 6 months
  if there is any inflammatory reaction, lost anterior chamber , cystoid macular edema

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eid, MD, Study Director — Minia University Hospital
Locations (1):
- Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramp K, Vick HP, Guthoff R. Transscleral diode laser contact cyclophotocoagulation in the treatment of different glaucomas, also as primary surgery. Graefes Arch Clin Exp Ophthalmol. 2002 Sep;240(9):698-703. doi: 10.1007/s00417-002-0508-5. Epub 2002 Aug 1. PMID 12271364
- [Background] Egbert PR, Fiadoyor S, Budenz DL, Dadzie P, Byrd S. Diode laser transscleral cyclophotocoagulation as a primary surgical treatment for primary open-angle glaucoma. Arch Ophthalmol. 2001 Mar;119(3):345-50. doi: 10.1001/archopht.119.3.345. PMID 11231767
- [Background] Quigley HA. The Need for Rigor in Evaluating Micropulse and Other New Procedures. Ophthalmol Glaucoma. 2020 May-Jun;3(3):171-173. doi: 10.1016/j.ogla.2020.04.004. No abstract available. PMID 32672611
- [Background] Sheheitli H, Persad PJ, Feuer WJ, Sayed MS, Lee RK. Treatment Outcomes of Primary Transscleral Cyclophotocoagulation. Ophthalmol Glaucoma. 2021 Sep-Oct;4(5):472-481. doi: 10.1016/j.ogla.2020.12.014. Epub 2021 Jan 8. PMID 33429109
- [Background] Khodeiry MM, Liu X, Lee RK. Clinical outcomes of slow-coagulation continuous-wave transscleral cyclophotocoagulation laser for treatment of glaucoma. Curr Opin Ophthalmol. 2022 May 1;33(3):237-242. doi: 10.1097/ICU.0000000000000837. Epub 2022 Feb 23. PMID 35200163
- [Background] Duerr ER, Sayed MS, Moster S, Holley T, Peiyao J, Vanner EA, Lee RK. Transscleral Diode Laser Cyclophotocoagulation: A Comparison of Slow Coagulation and Standard Coagulation Techniques. Ophthalmol Glaucoma. 2018 Sep-Oct;1(2):115-122. doi: 10.1016/j.ogla.2018.08.007. Epub 2018 Aug 25. PMID 32632402
- [Background] Moussa K, Feinstein M, Pekmezci M, Lee JH, Bloomer M, Oldenburg C, Sun Z, Lee RK, Ying GS, Han Y. Histologic Changes Following Continuous Wave and Micropulse Transscleral Cyclophotocoagulation: A Randomized Comparative Study. Transl Vis Sci Technol. 2020 Apr 28;9(5):22. doi: 10.1167/tvst.9.5.22. eCollection 2020 Apr. PMID 32821494
- [Background] Conlon R, Saheb H, Ahmed II. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017 Feb;52(1):114-124. doi: 10.1016/j.jcjo.2016.07.013. Epub 2016 Nov 17. PMID 28237137
- [Background] Oh LJ, Wong E, Lam J, Clement CI. Comparison of bleb morphology between trabeculectomy and deep sclerectomy using a clinical grading scale and anterior segment optical coherence tomography. Clin Exp Ophthalmol. 2017 Sep;45(7):701-707. doi: 10.1111/ceo.12953. Epub 2017 May 9. PMID 28371125
- [Background] Takihara Y, Inatani M, Seto T, Iwao K, Iwao M, Inoue T, Kasaoka N, Murakami A, Futa R, Tanihara H. Trabeculectomy with mitomycin for open-angle glaucoma in phakic vs pseudophakic eyes after phacoemulsification. Arch Ophthalmol. 2011 Feb;129(2):152-7. doi: 10.1001/archophthalmol.2010.348. PMID 21320958
- [Background] Correia Barbosa R, Goncalves R, Bastos R, Alves Pereira S, Basto R, Viana AR, Tenedorio P. Trabeculectomy Vs Non-penetrating Deep Sclerectomy for the Surgical Treatment of Open-Angle Glaucoma: A Long-Term Report of 201 Eyes. Clin Ophthalmol. 2023 Jun 6;17:1619-1627. doi: 10.2147/OPTH.S405837. eCollection 2023. PMID 37304331
- [Background] Pantalon A, Feraru C, Tarcoveanu F, Chiselita D. Success of Primary Trabeculectomy in Advanced Open Angle Glaucoma. Clin Ophthalmol. 2021 May 27;15:2219-2229. doi: 10.2147/OPTH.S308228. eCollection 2021. PMID 34079219
- [Background] Weinreb RN, Aung T, Medeiros FA. The pathophysiology and treatment of glaucoma: a review. JAMA. 2014 May 14;311(18):1901-11. doi: 10.1001/jama.2014.3192. PMID 24825645
- [Background] Zhang N, Wang J, Li Y, Jiang B. Prevalence of primary open angle glaucoma in the last 20 years: a meta-analysis and systematic review. Sci Rep. 2021 Jul 2;11(1):13762. doi: 10.1038/s41598-021-92971-w. PMID 34215769
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Melik Parsadaniantz S, Reaux-le Goazigo A, Sapienza A, Habas C, Baudouin C. Glaucoma: A Degenerative Optic Neuropathy Related to Neuroinflammation? Cells. 2020 Feb 25;9(3):535. doi: 10.3390/cells9030535. PMID 32106630

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT07152132/Prot_SAP_000.pdf